CLINICAL TRIAL: NCT06524089
Title: Pilates Versus Eccentric Exercises in Chronic Low Back Pain With Multiple Sclerosis
Brief Title: Pilates Versus Eccentric Exercises on Multiple Sclerosis
Acronym: MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Karima Abdelaty Hassan, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PILATES 2024
Record Dates: First submitted 2024-07-22; First posted 2024-07-29 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis
Keywords: Pilates; eccentric; multiple sclerosis; low back pain
MeSH Terms: conditions — Multiple Sclerosis; Low Back Pain

STUDY DESIGN:
Intervention Model Description: Parallel group prospective randomized clinical trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates (Experimental): Fifteen patients will receive Pilates exercises
  Interventions: Other: Pilate training
- eccentric (Experimental): Fifteen patients will receives eccentric training
  Interventions: Other: eccentric training

INTERVENTIONS:
Other: Pilate training — Pilates based training exercises group will perform Pilates divided into two levels (beginner and intermediate). Each level will last for six sessions.
  Arms: Pilates
Other: eccentric training — eccentric trunk training exercises group:The course of the intervention period is 12 sessions total, exercises performed for two to three sets with 10 to 15 repetitions each set and 2 min rest between each set
  Arms: eccentric

SUMMARY:
This study aims to determine whether Pilates-based stability or eccentric training is more effective for patients with multiple sclerosis(MS) with chronic non-specific low back pain(NSLBP).

DETAILED DESCRIPTION:
Thirty adult patients with multiple sclerosis with chronic NSLBP verified diagnosis of MS by a specialized neurologist will be questioned and screened according to inclusion and exclusion criteria.

Patients were randomly allocated to one of two groups: (Pilates or Eccentric). Every individual in both groups will be examined before and after the 6-week treatment program.

The handheld dynamometer assessed isometric trunk flexion and extension strength Pain intensity by casual analog scale (VAS). The Trunk Impairment Scale (TIS) evaluates static and dynamic sitting balance and trunk coordination in a seated position.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18 to 40 years.
* Relapsing-remitting free for at least 90 days before testing.

Exclusion Criteria:

* Having a neurologic disease other than MS.
* A relapse within 3 months.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-07-30 (Actual); Primary Completion 2025-03-02 (Actual); Study Completion 2025-03-02 (Actual)

PRIMARY OUTCOMES:
pain intensity | At baseline and after 6 week
  VAS for measuring pain severity
Function | At baseline and after 6 week
  The Trunk impairment scale (TIS) The static subscale investigates: (1) the ability of the subject to maintain a sitting position with feet supported; (2) the ability to maintain a sitting position while the legs are passively crossed, and (3) the ability to maintain a sitting position when the subject crosses the legs actively. The dynamic subscale contains items on lateral flexion of the trunk and unilateral lifting of the hip. To assess the coordination of the trunk, the subject is asked to rotate the upper or lower part of his or her trunk 6 times, initiating the movements either from the shoulder girdle or from the pelvic girdle, respectively. For each item, a 2-, 3- or 4- point ordinal scale is used. On the static and dynamic sitting balance and coordination subscales the maximal scores that can be attained are 7, 10 and 6 points. Therefore, TIS ranges between 0 for a minimal performance to 23 for a perfect performance.

SECONDARY OUTCOMES:
back muscle strength | At baseline and after 6 week
  Handheld dynamometer measuring isometric trunk muscle strength

CONTACTS AND LOCATIONS:
Overall Officials: Karima A Hassan, Study Director — Cairo University
Locations (1):
- Cairo university hospital, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duff WRD, Andrushko JW, Renshaw DW, Chilibeck PD, Farthing JP, Danielson J, Evans CD. Impact of Pilates Exercise in Multiple Sclerosis: A Randomized Controlled Trial. Int J MS Care. 2018 Mar-Apr;20(2):92-100. doi: 10.7224/1537-2073.2017-066. PMID 29670495
- [Background] Demaneuf T, Aitken Z, Karahalios A, Leong TI, De Livera AM, Jelinek GA, Weiland TJ, Marck CH. Effectiveness of Exercise Interventions for Pain Reduction in People With Multiple Sclerosis: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Arch Phys Med Rehabil. 2019 Jan;100(1):128-139. doi: 10.1016/j.apmr.2018.08.178. Epub 2018 Sep 19. PMID 30240593